CLINICAL TRIAL: NCT05040646
Title: Study Protocol - The Development of a Novel Patient Reported Outcomes Measure Committed to the Watch-and-wait Program for Rectal Cancer: An International Delphi Study Protocol
Brief Title: The Development of a Patient Reported Outcomes Measure Committed to the Watch-and-wait Program for Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-2805
Record Dates: First submitted 2021-06-29; First posted 2021-09-10 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2021-06

CONDITIONS: Rectal Cancer
Keywords: Watch-and-wait; Organ-preserving treatment method; Functional outcomes; Patient reported outcome measures; Quality of life; Delphi exercise
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients who follow the watch-and-wait program for rectal cancer.
  Interventions: Other: Delphi exercise
- Experts: Surgeons, radiotherapists, medical oncologist and other medical personnel who are involved in the treatment of rectal cancer and the watch-and-wait program.
  Interventions: Other: Delphi exercise

INTERVENTIONS:
Other: Delphi exercise — During the Delphi exercise both patients and experts will participate in two anonymous online survey rounds where different items/outcomes will be presented that are possibly related to rectal cancer and the W&W program. Both groups are asked to rate each item on a 9 point likert scale with respect to the importancy of the item.
  After the two subsequent rounds, participants will be invited to attend a consensus meeting, where final consensus about the most important outcomes will be reached.

SUMMARY:
The purpose of this study to develop an international tool that can be used to assess burden of disease in patients enrolled in the W&W program for rectal cancer

DETAILED DESCRIPTION:
The watch-and-wait (W&W) strategy in rectal cancer is a organ-sparing treatment option, where patients with a clinical complete response (cCR) after neoadjuvant chemo(radio)therapy, do not undergo surgery but instead follow a strict follow-up scheme. The goal of the W&W strategy is to preserve the rectum and thereby retain functional outcomes (FO) (e.g. gastro-intestinal, urinary, sexual) and improve quality of life (QoL).

Patient Reported Outcome Measures (PROMs) reflect the patients' evaluation of their symptoms, FO and QoL. In the W&W program various PROMs (e.g. EORTC-CR29/C30, LARS, SF-36) are used to assess the these different outcomes. However, most of the PROMs used are developed and validated in a surgical patient group. So the relevance and usefulness of these PROMs may be limited in W&W patients.

For use in clinical practice, a short PROM would support follow-up care as it provides a clear overview of the problems W&W patients experience.

This paper describes the protocol for the development of an international tool that can be used to assess burden of disease in patients enrolled in the W&W program for rectal cancer. We will use the Delphi methodology to reach consensus about items that should be included in the novel tool. The aim of this tool is to improve direct patient care during the entire Watch-and-Wait program.

ELIGIBILITY:
Inclusion Criteria:

* Patients have to be treated with neoadjuvant (chemo)radiotherapy
* Patients are included into the Watch-and-Wait program
* Experts involved in the treatment of rectal cancer
* Experts involved in the Watch-and-Wait program

Exclusion Criteria:

* Regrowth of disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of both patients and experts (surgeons, radiotherapist, medical oncologist and other medical personnel) who are involved in the watch-and-wait program for rectal cancer
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Consensus in / Important outcome | between 3 months and 5 years of follow up
  >70% of the participants in each panel rating the outcome '7-9' OR <70% of the clinicians and (clinical) researchers rating the outcome '7-9' but an average patient rating of >7
Consensus in / No important outcome | between 3 months and 5 years of follow up
  <70% of the clinicians and (clinical) researchers rating the outcome '7-9' AND an average patient rating of <7

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Breukink, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht UMC, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Greenhalgh J, Gooding K, Gibbons E, Dalkin S, Wright J, Valderas J, Black N. How do patient reported outcome measures (PROMs) support clinician-patient communication and patient care? A realist synthesis. J Patient Rep Outcomes. 2018 Sep 15;2:42. doi: 10.1186/s41687-018-0061-6. eCollection 2018 Dec. PMID 30294712
- [Background] Ishaque S, Karnon J, Chen G, Nair R, Salter AB. A systematic review of randomised controlled trials evaluating the use of patient-reported outcome measures (PROMs). Qual Life Res. 2019 Mar;28(3):567-592. doi: 10.1007/s11136-018-2016-z. Epub 2018 Oct 3. PMID 30284183
- [Background] Black N. Patient reported outcome measures could help transform healthcare. BMJ. 2013 Jan 28;346:f167. doi: 10.1136/bmj.f167. PMID 23358487
- [Background] Edwards P, Roberts I, Clarke M, DiGuiseppi C, Pratap S, Wentz R, Kwan I. Increasing response rates to postal questionnaires: systematic review. BMJ. 2002 May 18;324(7347):1183. doi: 10.1136/bmj.324.7347.1183. PMID 12016181
- [Background] Maas M, Beets-Tan RG, Lambregts DM, Lammering G, Nelemans PJ, Engelen SM, van Dam RM, Jansen RL, Sosef M, Leijtens JW, Hulsewe KW, Buijsen J, Beets GL. Wait-and-see policy for clinical complete responders after chemoradiation for rectal cancer. J Clin Oncol. 2011 Dec 10;29(35):4633-40. doi: 10.1200/JCO.2011.37.7176. Epub 2011 Nov 7. PMID 22067400
- [Background] van der Valk MJM, Hilling DE, Bastiaannet E, Meershoek-Klein Kranenbarg E, Beets GL, Figueiredo NL, Habr-Gama A, Perez RO, Renehan AG, van de Velde CJH; IWWD Consortium. Long-term outcomes of clinical complete responders after neoadjuvant treatment for rectal cancer in the International Watch & Wait Database (IWWD): an international multicentre registry study. Lancet. 2018 Jun 23;391(10139):2537-2545. doi: 10.1016/S0140-6736(18)31078-X. PMID 29976470
- [Background] Habr-Gama A, Sao Juliao GP, Fernandez LM, Vailati BB, Andrade A, Araujo SEA, Gama-Rodrigues J, Perez RO. Achieving a Complete Clinical Response After Neoadjuvant Chemoradiation That Does Not Require Surgical Resection: It May Take Longer Than You Think! Dis Colon Rectum. 2019 Jul;62(7):802-808. doi: 10.1097/DCR.0000000000001338. PMID 31188180
- [Background] Hsu, C. and B. Sandford, The Delphi technique: making sense of consensus-Practical assessment, research & evaluation. Pract Assessment. Res Eval, 2007. 12.